CLINICAL TRIAL: NCT01891500
Title: Effect of Early iNO on Oxidative Stress, Vascular Tone and Inflammation in Term and Late-Preterm Infants With Hypoxic Respiratory Failure
Brief Title: Early iNO for Oxidative Stress, Vascular Tone and Inflammation in Babies With Hypoxic Respiratory Failure
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficult to identify subjects who meet enrollment criteria.
Sponsor: University of Florida (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB201400791; 00089105 (Other: RAC); OCR17867 (Other: Universiy of Florida)
Record Dates: First submitted 2013-06-19; First posted 2013-07-03 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Persistent Fetal Circulation Syndrome; Hypertension, Pulmonary, of Newborn, Persistent; Persistent Pulmonary Hypertension of Newborn
Keywords: Persistent Fetal Circulation Syndrome; Infant, Newborn; Nitric Oxide; Oxidative Stress; Endothelin 1; Vascular Endothelial Growth Factor
MeSH Terms: conditions — Persistent Fetal Circulation Syndrome | interventions — Endothelium-Dependent Relaxing Factors; Nitrogen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Early inhaled nitric oxide (Experimental): Patients randomized to receive iNO at OI 10-15.
  Interventions: Drug: Inhaled nitric oxide
- Bioinert inhaled gas (nitrogen gas) (Placebo Comparator): Patients randomized to bioinert inhaled gas at OI 10-15.
  Interventions: Drug: Nitrogen Gas
- Crossover iNO (Active Comparator): Patients who deteriorate (OI >20 on two consecutive blood gases) will be unblinded. If they are receiving placebo gas, they will be started on iNO and make up the crossover cohort.
  Interventions: Drug: Crossover iNO

INTERVENTIONS:
Drug: Inhaled nitric oxide — Drug is initiated at 20ppm. Patients randomized to receive iNO at OI 10-15.
  Other Names: INOmax
  Arms: Early inhaled nitric oxide
Drug: Nitrogen Gas — Placebo gas (bioinert), Patients randomized to bioinert inhaled gas at OI 10-15.
  Other Names: bioinert
  Arms: Bioinert inhaled gas (nitrogen gas)
Drug: Crossover iNO — Patients who deteriorate (OI >20 on two consecutive blood gases) will be unblinded. If they are receiving placebo gas, they will be started on iNO and make up the crossover cohort.
  Other Names: bioinert; INOmax
  Arms: Crossover iNO

SUMMARY:
The investigators in this study are concerned about the harmful effects of oxygen exposure in newborn infants, particularly at high concentrations. Inhaled nitric oxide (iNO) is an FDA approved drug for the treatment of hypoxic respiratory failure (HRF) in term and late-preterm babies greater than 34 weeks gestation. Hypoxic respiratory failure occurs when a patient's lungs cannot get enough oxygen into their bloodstream. This condition is traditionally treated with high concentrations of oxygen and most often requires the patient be placed on a ventilator (breathing machine). The administration of inhaled nitric oxygen directly into the lungs often improves blood oxygen levels and allows caretakers to reduce the amount of oxygen given to the baby. The purpose of this research study is to evaluate if giving the inhaled nitric oxide earlier in the course of disease improves the effectiveness of the drug, reduces the amount of cellular injury from oxygen exposure, and decreases the total amount of time a patient requires supplemental oxygen. This study uses an FDA approved drug in a new manner.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≥ 35 weeks gestation
* Age of life ≤ 48 hours
* Diagnosis of hypoxic respiratory failure (HRF) as defined by a post-ductal SaO2 ≤90% in ≥50% oxygen with a PEEP of ≥ 6cm or an oxygenation index (OI) ≥ 10 but ≤ 15 when mean airway pressure and PaO2 are known.
* Mothers (ages 18 - 65) of eligible subjects for additional data collection

Exclusion Criteria:

* Gestational age < 35 weeks gestation.
* Post-natal age > 48 hours.
* Previous treatment with 100% oxygen for longer than 4 hours.
* Confirmed congenital diaphragmatic hernia.
* Suspected or confirmed congenital airway or pulmonary anomaly.
* Suspected or confirmed chromosomal anomaly or genetic aberration, with the exception of patients with trisomy 21 who do not have complex congenital heart disease.
* Infants with pneumothorax as the primary cause of their HRF.
* Infants with confirmed complex congenital heart disease.

Ages: 30 Minutes to 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-19 (Actual)

PRIMARY OUTCOMES:
Biomarkers of oxidative injury. | Urine samples will be collected upon enrollment and then at specific time points within the first 48 hours of study intervention to compare the change in biomarker concentrations from baseline up to hour 48.
  Early administration of iNO to infants with HRF will result in reduced hyperoxia-mediated oxidative injury as measured by known biomarkers of oxygen free radical injury, including malondialdehyde and 8-hydroxy-2'-deoxyguanosine.

SECONDARY OUTCOMES:
Responsiveness to study treatment. | Arterial oxygen concentration will be measured upon enrollment and at specific time points in the first 36 hours of study intervention to compare the change in arterial oxygen concentration from baseline up to hour 36.
  Earlier administration of iNO to infants with HRF/PPHN (persistent pulmonary hypertension of the newborn) will lessen reactive oxygen species formation resulting in improved responsiveness to the drug as measured by the initial changes in arterial oxygen concentration after administration of the drug.
Expression of endothelin-1. | Concentration of endothelin-1 will be measured upon enrollment and at specific time points in the first 36 hours of study intervention to compare the change in concentration from baseline up to hour 36.
  Earlier treatment with iNO may potentiate pulmonary vasodilation by modulating endothelin-1 expression.
Markers of inflammation. | Concentrations of pro and anti-inflammatory markers will be measured upon enrollment and at specific time points in the first 36 hours of study intervention to compare the change in concentrations from baseline up to hour 36.
  Early iNO may up-regulate production of endogenous anti-inflammatory eicosanoids such as PGE2 (prostaglandin E2). Additionally, avoidance of hyperoxia in these patients may mitigate pro-inflammatory cytokines known to potentiate lung injury.
Duration of oxygen treatment. | Participants will be followed for the duration of their hospital stay, with an expected average stay of 4 weeks.
  Early administration of iNO to infants with HRF will result in at least a 15% reduction in total days of oxygen therapy.
Expression of VEGF (vascular endothelial growth factor). | Concentration of VEGF will be measured upon enrollment and at specific time points in the first 36 hours of study intervention to compare the change in concentration from baseline up to hour 36.
  Earlier treatment with iNO may potentiate pulmonary vasodilation by preventing hyperoxic down regulation of VEGF.

CONTACTS AND LOCATIONS:
Overall Officials: Catalina Bazacliu, MD, Principal Investigator — University of Florida
Locations (1):
- Shands Hospital at the University of Florida, Gainesville, Florida, United States